CLINICAL TRIAL: NCT02201303
Title: A Single-Center In Vitro Study to Evaluate GSK1325756 Inhibition of CD11b Cell Surface Expression in Healthy Adults and Respiratory Syncytial Virus-Infected Children <2 Years (200591)
Brief Title: Evaluation of Danirixin (GSK1325756) Inhibition of CD11b Cell Surface Expression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200591
Record Dates: First submitted 2014-01-09; First posted 2014-07-28 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Infections, Respiratory Syncytial Virus
Keywords: CD11b; Neutrophils; CXCL1; Danirixin; Respiratory Syncytial Virus; Children; CXCR2
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — danirixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Blood sample will be collected from the RSV-infected children <2 years and healthy adults participants. Escalating concentrations of CXCL1 will be added to whole blood in vitro and CD11b up regulation on peripheral blood neutrophils will be analyzed
  Interventions: Other: CXCL1
- Part 2 (Experimental): Blood sample will be collected from the RSV-infected children <2 years and healthy adults participants. Escalating concentrations of danirixin will be added to whole blood in vitro with a fixed concentration of CXCL1 to determine inhibition of CD11b expression on peripheral blood neutrophils
  Interventions: Drug: Danirixin; Other: CXCL1

INTERVENTIONS:
Drug: Danirixin — Powdered form for in-vitro administration to blood sample
  Arms: Part 2
Other: CXCL1 — Escalating concentrations of CXCL1 will be added to whole blood in vitro. A CXCL1/CD11b upregulation concentration response curve will determine the concentration to be used in Part 2.

SUMMARY:
This study is to determine danirixin (GSK1325756) concentrations required to inhibit neutrophil activation in blood obtained from Respiratory Syncytial Virus (RSV)-infected children <2 years and healthy adults. The study will evaluate differences in neutrophil activation between RSV-infected children <2 years and healthy adults with escalating concentrations of Chemokine (C-X-C motif) Ligand 1 (CXCL1) and danirixin to determine if RSV-infected children and adult neutrophils are similarly activated by CXCL1 and inhibited by danirixin. This study will guide dose prediction to inhibit specific percentages of neutrophils in future pediatric RSV-infection studies. This single-center, in vitro study will consist of 2 parts. Approximately 24 subjects will be enrolled, including 12 healthy adults and 12 RSV-infected children <2 years.

ELIGIBILITY:
Inclusion Criteria:

Healthy Adults

* Male/females aged between 18 and 64 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history and physical examination. A subject with a clinical abnormality parameter(s) which is not specifically listed in the inclusion or exclusion criteria, may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 45 kilograms (kg) and body mass index (BMI) within the range 18.5-32 kg/meter^2 (inclusive).
* A female subject is eligible to participate if she is not known to be pregnant by history or delivered within the past 3 months.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

RSV Infected Children

* Male/females aged <2 years, at the time of parent(s)/legal guardian(s) signing the informed consent.
* Healthy, except for current RSV-infection, as determined by a responsible and experienced physician, based on a medical evaluation including medical history and physical examination. A subject with a clinical abnormality parameter(s) which is not specifically listed in the inclusion or exclusion criteria, may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 3.5 kg
* Documented RSV-infection, either by RSV-antigen or RSV-PCR
* RSV-infection clinical symptom onset within 5 days of blood draw based on parent(s)/guardian(s) history.
* Parent(s)/legal guardian(s) of child capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

Healthy Adults

* Any clinical infection within the past 14 days per subject's history.
* Acute or chronic infectious/inflammatory diseases by history, including but not limited to, hepatitis B, hepatitis C, human immuno virus (HIV), inflammatory bowel disease, liver / biliary disease, pancreatitis, arthritis.
* Receiving systemic anti-inflammatory or immune modulating medications, including but not limited to, non-steroidal anti-inflammatory (NSAIDS) and glucocorticoids, within the past 14 days. All other medications are permitted.
* Any alcoholic beverage within 24 hours of blood collection and history of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Current smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Strenuous exercise within 48 hours prior to the blood collection.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to signing the informed consent in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

RSV Infected Children

* A Child in Care: A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. A child in care can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. A child in care does not include a child who is adopted or has an appointed legal guardian.
* Any clinical infection, besides current RSV infection, within the past 14 days per subject's history
* Acute or chronic infectious/inflammatory diseases by history, including but not limited to, hepatitis B, hepatitis C, HIV, liver / biliary disease, pancreatitis
* Receiving systemic anti-inflammatory or immune modulating medications, including but not limited to, NSAIDS and glucocorticoids, within the past 14 days. All other medications are permitted.
* Past medical history including prematurity <37 weeks, congenital heart disease, chronic lung disease, or immunodeficiency.
* Where participation in the study would result in withdrawal of blood or blood products in excess of 2 mL/kg for 24 hours before or after the study period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to parent(s)/guardian(s) signing the informed consent in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Max Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2015-07-02 (Actual)

PRIMARY OUTCOMES:
Percent inhibition of Chemokine Ligand (CXCL1)-induced Cluster of Differentiation 11b expression on peripheral blood neutrophils in RSV-infected children <2 years and healthy adults after in vitro incubation with escalating concentrations of danirixin | Day 1
  Blood (1.5 milliliter [mL]) will be collected from a peripheral vein via indwelling catheter or direct venepuncture. Escalating concentrations of danirixin (0.03-100 micromoles) will be added to whole blood in vitro with a fixed concentration of CXCL1 to determine inhibition of Cluster of Differentiation 11b (CD11b) expression on peripheral blood neutrophils analyzed by Fluorescence-Activated Cell sorting (FACs).

SECONDARY OUTCOMES:
CD11b upregulation on peripheral blood neutrophils in RSV-infected children <2 years and healthy adults after in vitro incubation with escalating concentrations of CXCL1 | Day 1
  Blood (1.0 mL) will be collected from a peripheral vein via indwelling catheter or direct venepuncture. Escalating concentrations of CXCL1 will be added to whole blood in vitro and CD11b upregulation on peripheral blood neutrophils will be analyzed by FACS
Differences in percent inhibition of CXCL1-induced CD11b expression on peripheral blood neutrophils in RSV-infected children <2 years and healthy adults after in vitro incubation with escalating concentrations of danirixin | Day 1
  Inhibition of CD11b upregulation will be evaluated to determine if there is a similar concentration-response relationship between healthy adults and RSV-infected children

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Syracuse, New York, United States

REFERENCES:
- See also: Results for study 200591 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200591?search=study&b'search_terms=200591'#rs